CLINICAL TRIAL: NCT03394885
Title: Atezolizumab in Combination With Neoadjuvant Chemotherapy and Interval Cytoreductive Surgery for Patients With Newly-Diagnosed Advanced-Stage Epithelial Ovarian Cancer
Brief Title: Atezolizumab With Neoadjuvant Chemotherapy for Patients With Newly-Diagnosed Advanced-Stage Ovarian Cancer
Acronym: AdORN
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Johns Hopkins University (Other); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00079313
Record Dates: First submitted 2017-11-29; First posted 2018-01-09 (Actual); Results first posted 2021-08-10 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Ovarian Cancer; Ovarian Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms | interventions — atezolizumab; Carboplatin; Paclitaxel; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Atezolizumab, Carboplatin, Paclitaxel (+Optional Bevacizumab) (Experimental): 1. Atezolizumab administered over 90 (± 15) minutes (for the first infusion, shortening to 60 (± 15) minutes and 30 ± 15) minutes for subsequent infusions as described below) followed by
  2. Paclitaxel 70-80mg/m2 IV administered over approximately one hour followed by
  3. Carboplatin IV administered over 15-30 minutes to achieve an initial target AUC of 5-6 mg/mL/Min (Calvert formula dosing).
  4. (Optional, Physician choice) Bevacizumab IV maintenance administered starting at cycle 5 of chemotherapy over 30-90 minutes. For those who receive bevacizumab, it will be given for a total duration of 16 cycles
  Interventions: Drug: Atezolizumab; Drug: Carboplatin; Drug: Paclitaxel; Drug: Bevacizumab

INTERVENTIONS:
Drug: Atezolizumab — 1200mg IV q3weeks
  Other Names: Tecentriq
Drug: Carboplatin — 5-6mg/ML IV q3 weeks
  Other Names: Paraplatin
Drug: Paclitaxel — 70-80 mg/m2 IV q1 week
  Other Names: Taxol
Drug: Bevacizumab — 15 mg/kg IV q3 weeks
  Other Names: Avastin

SUMMARY:
The main purpose of this study is to validate a safe dose of atezolizumab with dose-dense paclitaxel and carboplatin when utilized with neoadjuvant chemotherapy and interval cytoreductive surgery followed by maintenance atezolizumab in women with advanced ovarian cancer.

DETAILED DESCRIPTION:
This is a Phase IB non-randomized, single-arm, open-label study of atezolizumab in combination with primary NACT-ICS in patients with advanced-stage epithelial ovarian cancer. The target population is women with previously untreated epithelial ovarian cancer (including fallopian tube and primary peritoneal cancer) with advanced stage (FIGO III-IV) disease suitable for NACT and ICS. The following regimen will be administered every 3 weeks for 3 cycles prior to ICS, then for 3 cycles following ICS:

* Carboplatin AUC = 5 or 6 IV, D1 of each cycle
* Paclitaxel 70 to 80mg/m2 IV, over one hour, on D1, 8, 15 of each cycle
* Atezolizumab 1200mg IV D1 of each cycle of chemotherapy and will be continued as maintenance therapy every 3 weeks until there is a lack of clinical benefit, unacceptable toxicity, or a total duration of 18 months.
* Bevacizumab (15 mg/kg IV every 3 weeks) may be added at cycle 5 of chemotherapy as per FDA approval. Those who opt for bevacizumab will receive chemotherapy, atezolizumab, and bevacizumab for cycles 5 and 6 followed by atezolizumab and bevacizumab maintenance. Maintenance bevacizumab will be given for a total duration of 16 cycles. Patients who have completed chemotherapy may opt for bevacizumab in the maintenance setting only if the amendment to add bevacizumab was not approved before after they started maintenance therapy.
* Upon completion of concurrent chemotherapy and atezolizumab therapy, patients will commence maintenance treatment with atezolizumab + bevacizumab for a total of up 16 cycles of maintenance therapy (22 total cycles of atezolizumab, and 18 total cycles of bevacizumab).

Each cycle is 21 days in duration and will be administered in the outpatient setting. Limited individualized flexibility in dose assignment (as noted) is permitted per physician discretion in regards to advanced-stage disease, nutritional status, ascites, non-physiologic creatinine measurements, and other comorbidities.

Three cycles of NACT with atezolizumab will be administered every 3 weeks prior to ICS (occurring between cycles 3 and 4) followed by 3 additional cycles (cycles 4-6) of chemotherapy with atezolizumab. Surgery must be performed after the third course of chemotherapy as soon as nadir counts permit, but preferably within six weeks after the completion of the third chemotherapy cycle. Fourth cycle of chemotherapy is to be administered as soon as possible, but preferably no more than six weeks after ICS.

Safety monitoring, including assessment for irAEs, will occur at each cycle and for 90 days after the last administration of atezolizumab or until start of next anti-cancer regimen, whichever occurs first. Image assessment by CT scan or MRI will be performed at baseline, prior to ICS to assess response, after completion of 6 cycles of chemotherapy with atezolizumab to assess response at end of chemotherapy treatment, and as clinically indicated during the maintenance phase and after completion of study treatment to assess PFS. Disease progression/recurrence will be defined per RECIST criteria and will not include isolated asymptomatic progression on the basis of CA125 levels. Immune function analysis will be performed on blood and tumor samples obtained at two time points: 1. confirmatory biopsy prior to start of therapy and 2. ICS.

It is estimated that 40 patients will be enrolled at an accrual rate of 3-5 patients/month and followed for a median of 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form (ICF)
* Ability and willingness to comply with the requirements of the study protocol
* Age ≥ 18 years
* No prior treatment for primary advanced (stage III or IV) epithelial ovarian, fallopian tube, or primary peritoneal carcinoma
* Confirmation of diagnosis (by surgical excisional/incisional biopsy or imaging-guided core biopsy), and patients for whom the plan of management will include NACT followed by ICS. The decision to proceed with NACT will be at the treating physician's discretion and include patients with advanced stage disease considered at low likelihood for optimal cytoreduction with primary debulking surgery.
* All patients must have measurable disease per RECIST v1.1

Patients must meet the following criteria prior to initiation of study treatment:

* Histology consistent with high-grade epithelial ovarian cancer (excluding mucinous carcinoma, clear cell carcinoma, and carcinosarcoma)
* An adequate pre-treatment tumor biopsy is required to confirm histologic diagnosis. Acceptable options include laparoscopic biopsy or image-guided core needle biopsy (minimum of two cores). Fine needle aspiration (FNA) biopsy or cytology from ascites is not adequate.
* Adequate hematologic and end organ function, defined by the following laboratory results obtained within 14 days prior to the first study treatment
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1 or 2 (see Appendix 6)
* Peripheral neuropathy less than or equal to CTCAE Grade 1
* For female patients of childbearing potential, agreement (by patient) to use highly effective form(s) of contraception (i.e., one that results in a low failure rate [< 1% per year] when used consistently and correctly) and to continue its use at least until ICS or if ICS is not performed then 90 days post last dose of atezolizumab

Exclusion Criteria:

* Mucinous, low-grade histology, clear cell carcinoma, or carcinosarcoma
* Prior systemic chemotherapy for epithelial ovarian, fallopian tube, or primary peritoneal cancer.
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years. (Exceptions include basal cell or squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.)
* AEs from prior anticancer therapy that have not resolved to Grade ≤ 1 except for alopecia
* Bisphosphonate therapy for symptomatic hypercalcemia
* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; cirrhosis; fatty liver; and inherited liver disease
* Known primary central nervous system (CNS) malignancy or symptomatic CNS metastases
* Pregnancy, lactation, or breastfeeding
* Known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* Inability to comply with study and follow-up procedures
* History or risk of autoimmune disease, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Bell's palsy, Guillain-Barré syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis
* History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest computed tomography (CT) scan
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications
* History of HIV infection or active hepatitis B (chronic or acute) or hepatitis C infection
* Active tuberculosis
* Severe infections within 4 weeks prior to Cycle 1, Day 1, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
* Signs or symptoms of infection within 2 weeks prior to Cycle 1, Day 1
* Received oral or IV antibiotics within 2 weeks prior to Cycle 1, Day 1
* Administration of a live, attenuated vaccine within 4 weeks before Cycle 1, Day 1 or anticipation that such a live, attenuated vaccine will be required during the study
* Prior history of treatment with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, anti-CTLA4 or any other antibodies targeting co-stimulation or checkpoint pathways
* Treatment with systemic immunostimulatory agents (including but not limited to interferon [IFN] alpha or interleukin [IL]-2) within 6 weeks or five half-lives of the drug (whichever is shorter) prior to Cycle 1, Day 1
* Treatment with investigational agent within 4 weeks prior to Cycle 1, Day 1 (or within five half lives of the investigational product, whichever is longer)
* Treatment with systemic immunosuppressive medications (including but not limited to prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks prior to Cycle 1, Day 1
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Patients with prior allogeneic bone marrow transplantation or prior solid organ transplantation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2020-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angeles A Secord, MD, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Duke Cancer Institute, Durham, North Carolina
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Atezolizumab, Carboplatin, Paclitaxel (+Optional Bevacizumab): 1. Atezolizumab administered over 90 (± 15) minutes (for the first infusion, shortening to 60 (± 15) minutes and 30 ± 15) minutes for subsequent infusions as described below) followed by
  2. Paclitaxel 70-80mg/m2 IV administered over approximately one hour followed by
  3. Carboplatin IV administered over 15-30 minutes to achieve an initial target AUC of 5-6 mg/mL/Min (Calvert formula dosing).
  4. (Optional, Physician choice) Bevacizumab IV maintenance administered starting at cycle 5 of chemotherapy over 30-90 minutes. For those who receive bevacizumab, it will be given for a total duration of 16 cycles
  Atezolizumab: 1200mg IV q3weeks
  Carboplatin: 5-6mg/ML IV q3 weeks
  Paclitaxel: 70-80 mg/m2 IV q1 week
  Bevacizumab: 15 mg/kg IV q3 weeks
Period: Overall Study
Arm/Group | Atezolizumab, Carboplatin, Paclitaxel (+Optional Bevacizumab)
Started | 18
Completed | 3
Not Completed | 15
Not completed — Adverse Event | 4
Not completed — Lack of Efficacy | 1
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 8
Not completed — Alternative Therapy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Atezolizumab, Carboplatin, Paclitaxel (+Optional Bevacizumab)
Number analyzed (Participants) | 18
Age, Continuous [Median (Standard Deviation); unit: years] | 67.9 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 14
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety: Incidence of Post Chemotherapy Surgical Debulking
Description: The number of subjects able to undergo interval cytoreductive surgery will be utilized as a measure of safety regarding the initial dosing of atezolizumab.
Time Frame: 9 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab, Carboplatin, Paclitaxel (+Optional Bevacizumab)
Number analyzed (Participants) | 18
Participants | 15
Statistical Analysis 1: Comparison: Atezolizumab, Carboplatin, Paclitaxel (+Optional Bevacizumab); Test type: Other; Exact Binomial Confidence Interval = 83, 95% CI 2-sided [66 to 100]

2. Primary Outcome: Safety: Incidence of Treatment Emergent Adverse Events
Description: The number of adverse events experienced while receiving study drugs will be utilized to assess safety of atezolizumab.
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab, Carboplatin, Paclitaxel (+Optional Bevacizumab)
Number analyzed (Participants) | 18
Participants
  None (Grade 0) | 1
  Mild (Grade 1) | 2
  Moderate (Grade 2) | 9
  Severe (Grade 3) | 4
  Life Threatening (Grade 4) | 2
  Lethal (Grade 5) | 0

3. Primary Outcome: Safety: Dose Intensity
Description: Percentage of planned doses of atezolizumab received at each cycle (21 day period) will be utilized as a measure of safety and tolerability for each subject.
Time Frame: Cycles 1-6,18 months total
Population: Participants planned to receive atezolizumab at each cycle.
Measure: Number; unit: percentage of planned doses
Arm/Group | Atezolizumab, Carboplatin, Paclitaxel (+Optional Bevacizumab)
Number analyzed (Participants) | 18
percentage of planned doses
  Cycle 1 | 100.0
  Cycle 2: number analyzed (Participants) | 16
  Cycle 2 | 81.3
  Cycle 3: number analyzed (Participants) | 15
  Cycle 3 | 93.3
  Cycle 4: number analyzed (Participants) | 15
  Cycle 4 | 86.7
  Cycle 5: number analyzed (Participants) | 15
  Cycle 5 | 86.7
  Cycle 6: number analyzed (Participants) | 15
  Cycle 6 | 100.0

4. Primary Outcome: Safety: Incidence of Dose Modifications
Description: The number of dose modifications for atezolizumab at each cycle (21 day period) will be utilized as a measure of safety and tolerability for each subject. Dose modifications are defined as doses delayed, doses discontinued, or doses held.
Time Frame: Cycles 1-6,18 months total
Population: Participants who received atezolizumab at each cycle.
Measure: Number; unit: dose modifications
Arm/Group | Atezolizumab, Carboplatin, Paclitaxel (+Optional Bevacizumab)
Number analyzed (Participants) | 18
dose modifications
  Cycle 1 | 0
  Cycle 2: number analyzed (Participants) | 16
  Cycle 2 | 3
  Cycle 3: number analyzed (Participants) | 15
  Cycle 3 | 1
  Cycle 4: number analyzed (Participants) | 15
  Cycle 4 | 2
  Cycle 5: number analyzed (Participants) | 15
  Cycle 5 | 3
  Cycle 6: number analyzed (Participants) | 15
  Cycle 6 | 2

5. Secondary Outcome: Number of Participants With a Complete or Partial Response as Measured by RECIST (Response Evaluation Criteria in Solid Tumors)
Description: RECIST criteria will be utilized for subjects over the course of the study to measure their response to study drugs. A Complete Response (disappearance of all tumor lesions) or Partial Response (reduction of greater than 30% in total tumor size) is considered a response.
Time Frame: 18 months
Population: Five participants were not evaluable for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab, Carboplatin, Paclitaxel (+Optional Bevacizumab)
Number analyzed (Participants) | 13
Participants | 12

6. Secondary Outcome: Number of Participants With Pathologic Complete Remission
Description: Cytoreduction pathologic complete remission will be measured using RECIST (Response Evaluation Criteria in Solid Tumors) and immune-related response criteria.
Time Frame: 9 weeks
Population: Three participants were not evaluable for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab, Carboplatin, Paclitaxel (+Optional Bevacizumab)
Number analyzed (Participants) | 15
Participants | 0

7. Secondary Outcome: Progression Free Survival Rate
Description: All patients will be evaluated for progression free survival from the date of first treatment to the date of first observation of progressive disease or death due to any cause or will be stopped at date of last follow-up for those still alive without disease progression. 18-month progression free survival rate as estimated by Kaplan-Meier method.
Time Frame: 18 months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Atezolizumab, Carboplatin, Paclitaxel (+Optional Bevacizumab)
Number analyzed (Participants) | 18
proportion of participants | 0.65 [0.26 to 0.92]

8. Secondary Outcome: Overall Survival Rate
Description: All patients will be evaluated for overall survival from the date of first treatment on protocol to the date of death due to any cause and will be stopped at date of last follow-up for those still alive.18-month overall survival rate as estimated by Kaplan-Meier method.
Time Frame: 18 months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Atezolizumab, Carboplatin, Paclitaxel (+Optional Bevacizumab)
Number analyzed (Participants) | 18
proportion of participants | 0.93 [0.82 to 1.00]

9. Other Pre Specified Outcome: Translational: PD-L1 Expression
Description: Analyzing changes in PD-L1 expression measured based on: immunohistochemistry after treatment with atezolizumab, association with BRCA mutation status, tumor mutation profile (next generation sequencing), and progression free survival.
Time Frame: 18 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Translational: Tumor Infiltrating Lymphocytes
Description: Analyzing changes in tumor infiltrating lymphocytes expression based on: immunohistochemistry after treatment with atezolizumab, association with BRCA mutation status, tumor mutation profile (next generation sequencing) and progression free survival.
Time Frame: 18 months
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Translational: Immune Checkpoint Receptors
Description: Analyzing changes in immune checkpoint receptor expression based on: flow cytometry after treatment with atezolizumab, association with BRCA mutation status, tumor mutation profile (next generation sequencing) and progression free survival.
Time Frame: 18 months
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Translational: Fold Change in Cytokine Expression
Description: Analyzing changes in cytokine expression based on: ELISA (enzyme-linked immunosorbent assay) after treatment with atezolizumab, association with BRCA mutation status, tumor mutation profile (next generation sequencing) and progression free survival.
Time Frame: Baseline, 18 months
Population: Data not collected on 4 participants.
Measure: Median (Full Range); unit: Fold change
Arm/Group | Atezolizumab, Carboplatin, Paclitaxel (+Optional Bevacizumab)
Number analyzed (Participants) | 14
Fold change
  CXCL10 Fold Change | 0.7 [0.2 to 3.8]
  INFgamma Fold Change | 0.8 [0.0 to 6.0]
  IL10 Fold Change | 0.9 [0.2 to 1.5]
  IL12p70 Fold Change | 1.4 [0.0 to 13.5]
  IL1b Fold Change | 0.9 [0.2 to 16.5]
  IL2RA Fold Change | 1.1 [0.4 to 2.8]
  IL6 Fold Change | 0.4 [0.0 to 5.6]
  TNFalpha Fold Change | 0.8 [0.2 to 1.9]
  TIM3 Fold Change | 1.0 [0.6 to 2.3]

13. Other Pre Specified Outcome: Translational: Gene Expression Profiles
Description: Analyzing changes in gene expression profiles based on: RNA sequencing after treatment with atezolizumab, association with BRCA mutation status, tumor mutation profile (next generation sequencing) and progression free survival.
Time Frame: 18 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Atezolizumab, Carboplatin, Paclitaxel (+Optional Bevacizumab)
All-Cause Mortality (participants affected / at risk) | 1/18
Serious Adverse Events (participants affected / at risk) | 4/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Atezolizumab, Carboplatin, Paclitaxel (+Optional Bevacizumab) (N=18)
Infections and infestations - Other: MRSA (Infections and infestations) | 1
Neutrophil count decreased (Investigations) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Thromboembolic event (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Atezolizumab, Carboplatin, Paclitaxel (+Optional Bevacizumab) (N=18)
Anemia (Blood and lymphatic system disorders) | 16
Leukocytosis (Blood and lymphatic system disorders) | 1
Mitral valve disease (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 4
Vertigo (Ear and labyrinth disorders) | 1
Hyperthyroidism (Endocrine disorders) | 4
Hypothyroidism (Endocrine disorders) | 3
Blurred vision (Eye disorders) | 1
Cataract (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 9
Ascites (Gastrointestinal disorders) | 2
Bloating (Gastrointestinal disorders) | 3
Colonic fistula (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 7
Diarrhea (Gastrointestinal disorders) | 12
Dry mouth (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 12
Oral pain (Gastrointestinal disorders) | 1
Rectal hemorrhage (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 5
Edema limbs (General disorders) | 6
Fatigue (General disorders) | 15
Fever (General disorders) | 1
Flu like symptoms (General disorders) | 2
General disorders and administration site conditions - Other, specify (General disorders) | 1
Malaise (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 5
Bacteremia (Infections and infestations) | 1
Bladder infection (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Eye infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Nail infection (Infections and infestations) | 1
Rhinitis infective (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 4
Bruising (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 7
Wound complication (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 5
Alkaline phosphatase increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 9
Blood bilirubin increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
CPK increased (Investigations) | 1
Creatinine increased (Investigations) | 2
Lymphocyte count decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 16
Platelet count decreased (Investigations) | 15
Thyroid stimulating hormone increased (Investigations) | 3
Weight gain (Investigations) | 1
Weight loss (Investigations) | 7
White blood cell decreased (Investigations) | 13
Anorexia (Metabolism and nutrition disorders) | 7
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 4
Hyperlipidemia (Metabolism and nutrition disorders) | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hyperphosphatemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 10
Hypocalcemia (Metabolism and nutrition disorders) | 10
Hypokalemia (Metabolism and nutrition disorders) | 9
Hypomagnesemia (Metabolism and nutrition disorders) | 10
Hyponatremia (Metabolism and nutrition disorders) | 8
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Myositis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 5
Headache (Nervous system disorders) | 6
Hypersomnia (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 14
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 3
Acute kidney injury (Renal and urinary disorders) | 1
Cystitis noninfective (Renal and urinary disorders) | 1
Glucosuria (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 2
Proteinuria (Renal and urinary disorders) | 3
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1
Urinary frequency (Renal and urinary disorders) | 4
Urinary urgency (Renal and urinary disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 2
Vaginal discharge (Reproductive system and breast disorders) | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 4
Vaginal inflammation (Reproductive system and breast disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 7
Dry skin (Skin and subcutaneous tissue disorders) | 7
Pruritus (Skin and subcutaneous tissue disorders) | 8
Rash acneiform (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2
Flushing (Vascular disorders) | 1
Hot flashes (Vascular disorders) | 1
Hypertension (Vascular disorders) | 7
Thromboembolic event (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-22): https://cdn.clinicaltrials.gov/large-docs/85/NCT03394885/Prot_SAP_000.pdf